CLINICAL TRIAL: NCT07004231
Title: Using Gout Buddy to Enhance Dietary Literacy and Gout Management-A Mixed Method Clinical Trial
Brief Title: Using Gout Buddy to Enhance Gout Management
Acronym: GOUTBuddy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SingHealth Polyclinics (Other)
Responsible Party: Principal Investigator, Tan Ngiap Chuan, Principal Investigator, SingHealth Polyclinics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-4476; 2024-4476 (Other: SINGHEALTH CENTRALISED INSTITUTIONAL REVIEW BOARD)
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Gout
Keywords: gout; dietary literacy; Artificial Intelligence; Chatbot; Primary care
MeSH Terms: conditions — Gout

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm using Gout Buddy (Experimental): Participants in the intervention group will receive usual care, including standard medical management and dietary counselling for gout. In addition, they will use the Gout Buddy chatbot (a prototype mobile application developed by HELF AI). The chatbot will be installed on their mobile phones (iOS or Android, 2020 models or newer) and requires a stable but standard mobile internet connectivity.
  Participants will download and enroll in Gout Buddy with the guidance of study team. The chatbot provides interactive support by allowing users to ask questions and receive daily tips and recommendations to help them manage their condition effectively.
  Notifications will be sent by Gout Buddy to the users' phones; these happen one to three times every day and mainly consist of daily tips related to better gout literacy and self-efficacy. The notifications are also useful conversation starters with users.
  Interventions: Other: GOUT Buddy, an AI chatbot
- Standard care (No Intervention): Participants in the control group will receive usual care, which includes standard medical management and dietary counselling for gout. They will also receive a pamphlet containing information on dietary management for gout.

INTERVENTIONS:
Other: GOUT Buddy, an AI chatbot — AI Chatbot ("GOUT Buddy") offers personalized gout education and awareness tailored to individual needs
  Arms: Intervention arm using Gout Buddy

SUMMARY:
Background: Dietary management is crucial for gout, but patients often lack adequate dietary literacy. However, patients often lack adequate dietary literacy and struggle to navigate complex dietary recommendations. Gout Buddy is an autonomous AI agent to offer personalized gout education and awareness tailored to individual needs. This study aims to evaluate the effectiveness and user experience of Gout Buddy, in improving dietary literacy and gout management.

Materials and methods: A two-arm RCT will randomize patients with gout to either the intervention (Gout Buddy) or control (standard care). Two study visits within 3-6 months will assess changes in dietary literacy and gout management behaviours. Qualitative interviews will be conducted with intervention arm participants and multidisciplinary care team members to explore their experiences with Gout Buddy till the point of data saturation.

Expected Outcomes: The current trial is expected to demonstrate the effectiveness of Gout Buddy in improving dietary literacy and gout management compared to standard care. Qualitative data will provide rich insights into user engagement, perceived benefits, challenges, and the feasibility of integrating the chatbot into routine gout management.

Significance: This study will provide evidence on the potential of AI chatbots to enhance gout self-management. The findings will inform the development and implementation of digital health tools for chronic disease management, potentially improving patient outcomes and reducing the burden of gout.

DETAILED DESCRIPTION:
Background and Rationale:

Gout is a chronic and progressive form of inflammatory arthritis characterized by the accumulation of urate crystals in the joints, leading to recurrent episodes of severe pain, redness, and swelling. It is primarily caused by hyperuricemia, a condition in which there is an excess of uric acid in the blood. Gout is more common in men and older adults and is often associated with comorbidities such as hypertension, diabetes, and cardiovascular disease.

A 2015 meta-analysis of global gout studies estimated a pooled prevalence of 0.6%, though with significant variation. [1] In mainland China, the prevalence of gout from 1998 to 2019 was 1.6%, and a local study from Singapore among Chinese individuals found that 4.1% had a history of physician-diagnosed gout. [2,3] Despite the availability of effective treatments, about one-third patients struggle with managing their condition.[4] Poor control can be attributed due to lack of understanding of gout's etiology, progression, and the importance of adherence to prescribed therapies. [5] Poor management of gout can result in frequent flare-ups, joint damage, and decreased quality of life.

Research indicates that patient education significantly impacts the successful management of gout. [6] However, traditional methods of patient education-such as pamphlets, infrequent consultations, and group sessions-often fall short in engaging patients and providing timely information tailored to their individual needs. [7,8] Additionally, these methods do not accommodate the continuous need for information that patients may have outside of clinic hours. Therefore, there is a need for innovative, accessible, and patient-centered educational tools that can bridge these gaps and empower patients to manage their gout more effectively.

Digital health interventions have emerged as a promising solution to these challenges. By leveraging technology, these interventions can provide continuous support, personalized information, and interactive educational content to patients. [9] Chatbots, in particular, have gained attention for their efficacy of health behaviour change among large and diverse population. [10] Chatbots can be particularly beneficial in chronic disease management, where ongoing patient education and engagement are critical. By providing instant access to reliable information and guidance, chatbots can help patients better understand their condition, adhere to treatment plans, and make informed decisions about their health.

Health Expert Language Framework (HELF) is a state-of-the-art AI-powered healthcare platform dedicated to advancing health and wellness education. Tailored for learners, educators, healthcare professionals, and researchers, HELF AI offers an immersive learning environment enriched by direct access to PubMed, a vast repository of the latest health literature. The platform elevates the educational experience by presenting detailed information and resources in a dynamic Question-Answer format, fostering a deeper understanding of health topics.

Building on this foundation, HELF AI can be further developed into a sophisticated, autonomous AI agent ("Gout Buddy") to offer personalized gout education and awareness tailored to individual needs. Given the challenges associated with gout management and the potential of digital health interventions, this study seeks to evaluate the effectiveness of the Gout Buddy as an intelligent patient companion, in improving dietary literacy of gout and adherence to its management, leveraging its AI capabilities to offer tailored educational support.

Study Objective:

1. To assess the effectiveness of the Gout Buddy in improving patients' dietary literacy of gout, adherence, and overall health outcomes
2. To explore the views, acceptance, and potential challenges associated with using the Gout Buddy among the participants and the multidisciplinary care team, including nurses, dietitians, and pharmacists.

The study will utilize the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance) to comprehensively evaluate the Gout Buddy intervention.

This study will employ a Sequential Explanatory mixed-methods design, incorporating both quantitative and qualitative approaches.

Quantitative phase: Two-arm randomized controlled trial (RCT) Arm 1: Usual care + Gout Buddy Arm 2: Usual care Qualitative phase: In-depth interviews will be conducted with participants who used the Gout Buddy, as well as the multidisciplinary care team (nurses, dietitians, and pharmacists) involved in patient care. These interviews will explore their experiences, views on the effectiveness of the chatbot, and any challenges they encountered. This will provide insights into the user experience and identify any barriers to effective implementation of Gout Buddy in managing patient care.

Recruitment and consent taking Participant recruitment Eligible patient participants will be identified through either screening from electronic medical records (EMR) or referred by the attending physicians to the study team. The study team will contact potential participants in-person or over phone to invite them to participate in the study and arrange a screening visit following which they will be recruited in-person during their regular clinic visits.

The study team will verify eligibility using a screening tool and written informed consent will be obtained in-person at the study site, in a quiet and separate room or space, ensuring privacy. Adequate time will be given to read the documents and questions, emphasizing the voluntary nature of participation and its independence from routine clinical care.

Participant withdrawal Participants may choose to withdraw from the study at any time without providing an explanation and this will not result in any punitive consequences.

Randomization Patient participants from each study site will be randomly allocated in a 1:1 ratio to one of the two arms in an open-label fashion, using computer-generated random numbers for simple randomization of subjects. The nature of the intervention makes impossible to blind patients and research team to participant allocation. The randomization sequence is written and kept in an opaque sealed envelope, which will be labelled with a serial number. The study team will open the sealed envelope once the patient has consented to participate and then will be assigned to the study arms accordingly.

Qualitative: In-depth interviews A semi-structured interview with retrospective probing, using an interview guide will be conducted among the participants who used the Gout Buddy, as well as with members of the multidisciplinary care team (nurses, dietitians, and pharmacists) involved in patient care till point of data saturation. Maximum variation sampling will be employed based on their age, ethnicity, and socioeconomic status. The session will be audio-recorded.

Follow-up Study participants will be followed up at their subsequent clinic visit, scheduled 3-6 months after enrolment, by a second assessor who is blinded to the intervention. If a participant does not return to the clinic within the study period, the follow up survey will be conducted via phone at a time convenient for them.

ELIGIBILITY:
Inclusion Criteria:

* Age > 21 years
* At least one serum uric acid > 360 μmol/L or an episode of acute gout attack within the last 18 months
* Able to read and speak English
* Access to an internet-enabled device compatible with Gout Buddy

Exclusion Criteria:

* Not a Singapore citizen or permanent resident
* Pregnant
* End-stage kidney disease or on renal replacement therapy
* Known terminal illness
* Visual and/or hearing impairment
* Cognitive impairment or mental illness
* Unable to provide informed consent
* Individuals who do not have a personal mobile device with internet access

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Food Frequency Questionnaire | through study completion, an average of 3 to 6 months
  Food Frequency Questionnaire-SF (FFQ-SF) is a limited checklist of foods and beverages with a frequency response section for subjects to report how often each item was consumed over a specified period of time. Changes in the frequency of consuming each food item will be compared to baseline consumption.
Dietary literacy about gout | through study completion, an average of 3 to 6 months
  Change in the scores using Dietary literacy about gout questionnaire; a newly developed questionnaire to assess patients' understanding of gout diet comprising 19 questions scored from a scale of 1-5: 1 (Strongly agree), 2 (agree), 3 (uncertain), 4 (disagree) and 5 (strongly disagree). A higher score indicates better understanding.
Medication adherence report scale- 5 items | through study completion, an average of 3 to 6 months
  Change in the scores using five item Medication Adherence Report Scale (MARS-5); MARS-5 score was calculated by summing the numeric score (range 1-5) from each question for out of 25 (range 5-25). A higher score indicates better adherence.
Health related quality of life (HRQoL) | through study completion, an average of 3 to 6 months
  Change in the scores using EQ-5D-5L questionnaire; The EQ-5D-5L tool comprises five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/ discomfort and anxiety/ depression. Each dimension has five response levels (no problems, slight problems, moderate problems, severe problems, unable to/ extreme problems). The proportion of patients reporting each level of problem on each dimension of the EQ-5D will be determined through study completion and compared. EQ VAS (Visual Analogue Scale) provides a quantitative measure of the patient's perception of their overall health. The EQ VAS records the respondent's overall current health on a vertical scale (0-100), where the endpoints are labelled '0-The worst health you can imagine' and '100-The best health you can imagine'.

SECONDARY OUTCOMES:
exploring the views, acceptance, and potential challenges associated with using the Gout Buddy | 3-6 months
  in-depth interview with the participants till point of data saturation

CONTACTS AND LOCATIONS:
Overall Officials: Ngiap Chuan Tan, MMed, Principal Investigator — SingHealth Polyclinics
Locations (1):
- SingHealth Polyclinics, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wijnands JM, Viechtbauer W, Thevissen K, Arts IC, Dagnelie PC, Stehouwer CD, van der Linden S, Boonen A. Determinants of the prevalence of gout in the general population: a systematic review and meta-regression. Eur J Epidemiol. 2015 Jan;30(1):19-33. doi: 10.1007/s10654-014-9927-y. Epub 2014 Jul 27. PMID 25064615
- [Background] Huang J, Ma ZF, Zhang Y, Wan Z, Li Y, Zhou H, Chu A, Lee YY. Geographical distribution of hyperuricemia in mainland China: a comprehensive systematic review and meta-analysis. Glob Health Res Policy. 2020 Nov 30;5(1):52. doi: 10.1186/s41256-020-00178-9. PMID 33292806
- [Background] Teng GG, Ang LW, Saag KG, Yu MC, Yuan JM, Koh WP. Mortality due to coronary heart disease and kidney disease among middle-aged and elderly men and women with gout in the Singapore Chinese Health Study. Ann Rheum Dis. 2012 Jun;71(6):924-8. doi: 10.1136/ard.2011.200523. Epub 2011 Dec 15. PMID 22172492
- [Background] Oka P, Chong WM, Ng DX, Aau WK, Tan NC. Epidemiology and risk factors associated with gout control among adult Asians: a real-world retrospective cohort study. Front Med (Lausanne). 2023 Sep 7;10:1253839. doi: 10.3389/fmed.2023.1253839. eCollection 2023. PMID 37746085
- [Background] Harrold LR, Mazor KM, Peterson D, Naz N, Firneno C, Yood RA. Patients' knowledge and beliefs concerning gout and its treatment: a population based study. BMC Musculoskelet Disord. 2012 Sep 21;13:180. doi: 10.1186/1471-2474-13-180. PMID 22995041
- [Background] Fields TR, Batterman A. How Can We Improve Disease Education in People with Gout? Curr Rheumatol Rep. 2018 Mar 8;20(3):12. doi: 10.1007/s11926-018-0720-x. PMID 29516200
- [Background] Bhattad PB, Pacifico L. Empowering Patients: Promoting Patient Education and Health Literacy. Cureus. 2022 Jul 27;14(7):e27336. doi: 10.7759/cureus.27336. eCollection 2022 Jul. PMID 36043002
- [Background] Hoving C, Visser A, Mullen PD, van den Borne B. A history of patient education by health professionals in Europe and North America: from authority to shared decision making education. Patient Educ Couns. 2010 Mar;78(3):275-81. doi: 10.1016/j.pec.2010.01.015. Epub 2010 Mar 1. PMID 20189746
- [Background] Kuwabara A, Su S, Krauss J. Utilizing Digital Health Technologies for Patient Education in Lifestyle Medicine. Am J Lifestyle Med. 2019 Dec 13;14(2):137-142. doi: 10.1177/1559827619892547. eCollection 2020 Mar-Apr. PMID 32231478
- [Background] Aggarwal A, Tam CC, Wu D, Li X, Qiao S. Artificial Intelligence-Based Chatbots for Promoting Health Behavioral Changes: Systematic Review. J Med Internet Res. 2023 Feb 24;25:e40789. doi: 10.2196/40789. PMID 36826990
- [Background] Serlachius A, Schache K, Kieser A, Arroll B, Petrie K, Dalbeth N. Association Between User Engagement of a Mobile Health App for Gout and Improvements in Self-Care Behaviors: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2019 Aug 13;7(8):e15021. doi: 10.2196/15021. PMID 31411147
- [Background] Rothenberg E, Strandhagen E, Samuelsson J, Ahlner F, Rydberg Sterner T, Skoog I, Lundberg CE. Relative Validity of a Short 15-Item Food Frequency Questionnaire Measuring Dietary Quality, by the Diet History Method. Nutrients. 2021 Oct 24;13(11):3754. doi: 10.3390/nu13113754. PMID 34836011